CLINICAL TRIAL: NCT01344486
Title: Peritoneal Cavity Conditioning During Laparoscopic Surgery Decreases Postoperative Pain, Inflammatory Reaction and Postoperative Adhesions
Brief Title: Peritoneal Cavity Conditioning Decreases Pain, Inflammation and Adhesions
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator no longer works fulltime at investigational site
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Jasper Verguts, MD, PhD, University Hospital, Gasthuisberg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: S52424
Record Dates: First submitted 2011-04-21; First posted 2011-04-29 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Endometriosis of the Cul-de-sac; Chocolate Cyst of Ovary; Fibroid/Myoma (Uterus/Cervix)
Keywords: women undergoing laparoscopic surgery
MeSH Terms: conditions — Endometriosis; Leiomyoma; Myoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full conditioing (Experimental): Intervention by alteration of laparoscopic gas with addition of oxygen and nitrous oxide, regulation of humidification and temperature (32°C), injection of 5mg Dexamethasone and application of Hyalobarrier Gel Endo (Nordic Pharma) at the surgical wound
  Interventions: Procedure: full conditioning
- carbon dioxide (Active Comparator): induction pneumoperitoneum with carbon dioxide 100%
  Interventions: Procedure: standard pneumoperitoneum

INTERVENTIONS:
Procedure: full conditioning — addition of 4% oxygen + 10% nitrous oxide to the pneumoperitoneum + humidification + temperature regulation at 32°C
  Arms: Full conditioing
Procedure: standard pneumoperitoneum — 100% carbon dioxide used for the pneumoperitoenum
  Arms: carbon dioxide

SUMMARY:
Full conditioning of the peritoneal cavity during laparoscopic surgery will decrease post-operative pain, inflammation and adhesion formation.

Full conditioning will decrease an inflammatory response of the peritoneum and decrease pain and adhesion formation.

DETAILED DESCRIPTION:
Randomized controlled trial (RCT) comparing carbon dioxide to full conditioning (addition of oxygen, nitrous oxide, humidification and temperature control, dexamethasone and Hyalobarrier gel) Women undergoing laparoscopy for endometriosis, myomectomy or adhesiolysis will be randomized to either group and will be compared for pain (VAS scores); inflammation (White blood cells, CRP) and adhesions scored by second look laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing laparoscopic excision of deep endometriosis (stratum 1), excision of endometrioma's (stratum 2) or excision of uterine myoma's (stratum 3) since this is severe surgery, associated with severe postoperative adhesions and since for most of these women fertility is important and hence the second look laparoscopy can be beneficial.
* Signed informed consent

Exclusion Criteria:

* women with a pre-existing condition increasing the risk of surgery such as clotting disorders, heart or lung impairment etc.-Any condition that might interfere with inflammatory parameters such as immunodeficiency, chronic inflammatory disease as Crohn's disease.
* Pregnancy
* Conditions associated with chronic pain as peripheral neuropathy, pathology of the vertebral column and osteo-articular disease. Conditions causing acute pain e.g. abdominal trauma
* a known allergic reaction to Hyalobarrier Gel Endo®
* A bowel lesion requiring a single or double layer suture. (given that for none of the anti-adhesion barriers safety has been proven following bowel lesions and suture)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
adhesion formation after laparoscopic surgery | 2 weeks after primary surgery
  second look laparoscopy to assess adhesions formed after initial surgery

SECONDARY OUTCOMES:
Post-operative pain | recorded until 3 days after surgery
  pain assessed by VAS scores
inflammation | recorded until 3 days after surgery
  bloodsamples to test for C reactive protein and white blood cells
time to first flatus and stool | recorded until 3 days after surgery
  patients will be asked when first flatus and first stool appeared. (measured as hours after surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Koninckx, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No